CLINICAL TRIAL: NCT06260865
Title: Prospective, Randomized, Controlled Confirmatory Clinical Investigation to Evaluate the Safety and Efficacy of a Multidisciplinary Digital Therapeutics in Patients with Patellofemoral Pain Syndrome
Brief Title: A Confirmatory Trial of Multidisciplinary Digital Therapeutics for Patellofemoral Pain Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EverEx Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-ETH-01K-CI02
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: PFPS; DTx; SaMD; MSK
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MORA Cure (Experimental): Participants randomly assigned to this arm will use the digital therapeutics, MORA Cure.
  Interventions: Device: MORA Cure
- Treatment as Usual (Active Comparator): Participants randomly assigned to this arm will receive their treatment as usual only.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Device: MORA Cure — MORA Cure (ETH-01K), developed by EverEx, Inc., is a digital therapeutics (S/W medical device) designed to provide multidisciplinary rehabilitation treatment, a combination of graded exercise therapy and cognitive behavioural therapy for patients with patellofemoral pain syndrome.
  Arms: MORA Cure
Other: Treatment as Usual — In the control group, education is delivered and self-exercise is recommended.
  Arms: Treatment as Usual

SUMMARY:
This randomized controlled confirmatory study will be evaluating an mobile application, MORA Cure (ETH-01K), owned by EverEx, Inc., to examine safety and effectiveness in individuals with patellofemoral pain syndrome.

DETAILED DESCRIPTION:
This randomized controlled confirmatory study will enroll 216 participants, where half will be randomly assigned to the digital therapeutics (S/W medical device), MORA Cure (n = 108), and half will be assigned to treatment as usual (TAU) (n = 108), to examine safety and effectiveness in individuals with patellofemoral pain syndrome. All subjects will be followed up in the study for a total of 12 weeks, 8-week courses of treatment with additional 4-week observation. The application provides multidisciplinary rehabilitation treatment, a combination of graded exercise therapy and cognitive behavioural therapy for patients with patellofemoral pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with peripatellar or posterior patellar pain in one or more knee joints for 3 months or longer
2. Patients with peripatellar or posterior patellar pain provoked by squatting
3. Patients who have pain provoked by 2 or more following activities: prolonged sitting, cycling, running, going up or down stairs, kneeling, compression of the patella, palpation of the patellar facets
4. Patients who signed a written informed consent form

Exclusion Criteria:

1. Patients with osteoarthritis which scored 3 or higher grade of the Kellgren-Lawrence scale
2. Patients diagnosed with a fracture or dislocation around the knee within the last 3 months
3. Patients who had knee surgery within the last 3 months
4. Patients diagnosed with patellar tendinitis based on imaging within 3 months
5. Patients taking narcotic pain medications for pain control
6. Patients taking or planning to take any medication that is a contraindication within the next 16 weeks at the time of screening
7. Patients who are pregnant
8. Patients currently participating in another clinical trial or have participated in another clinical trial within the past 3 months at the time of screening
9. Patients deemed unsuitable for this study by the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Usual pain severity assessed by the Visual Analogue Scale (VAS) | 8 weeks
  Differences in usual pain severity between groups after the intervention. VAS score will be measured from 0 (no pain) to 100 (worst pain imaginable).

SECONDARY OUTCOMES:
Usual pain severity assessed by the Visual Analogue Scale (VAS) | 4 weeks, 12 weeks
  Differences in usual pain severity between groups after the intervention. VAS score will be measured from 0 (no pain) to 100 (worst pain imaginable).
Worst pain severity assessed by the Visual Analogue Scale (VAS) | 4 weeks, 8 weeks, 12 weeks
  Differences in worst pain severity between groups after the intervention. VAS score will be measured from 0 (no pain) to 100 (worst pain imaginable).
Functional disability assessed by the Kujala Patellofemoral Scale | 4 weeks, 8 weeks, 12 weeks
  Differences in functional disability between groups. Kujala Patellofemoral Scale, also known as Anterior Knee Pain Scale, is a patient reported assessment of patellofemoral pain syndrome-specific functional limitations. It has 13 questions, and total score ranges from 0 to 100 (higher scores meaning better outcomes).
Health-related quality of life assessed by EuroQol five-dimensional (EQ-5D) | 4 weeks, 8 weeks, 12 weeks
  Differences in health-related quality of life between groups. It measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with three possible answers for each dimension (1=no problem, 2=moderate problem, 3=severe problem). The instrument also includes a visual analogue scale, which is numbered from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Assessment of mental health symptoms specific to depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | 4 weeks, 8 weeks, 12 weeks
  Differences in mental health symptoms between groups. The Patient Health Questionnaire-9 (PHQ-9) total score for the nine items ranges from 0 to 27 (higher scores indicating greater severity of depression).
Assessment of catastrophic thinking measured by Pain Catastrophizing Scale (PCS) | 4 weeks, 8 weeks, 12 weeks
  Differences in levels of catastrophic thinking between groups at 8, 12 weeks. The Pain Catastrophizing Scale (PCS) is a 13-item scale, with a total range of 0 to 52 (higher scores indicating higher amounts of pain catastrophizing).
Flexion and extension strength of knee | 4 weeks, 8 weeks, 12 weeks
  Flexion and extension strength of knee are measured using a Biodex isokinetic dynamometer (peak torque (Nm) and % decrease in torque).
Treatment adherence | 4 weeks, 8 weeks, 12 weeks
  Treatment adherence of each group, defined as percentage of days taking treament properly out of all days

CONTACTS AND LOCATIONS:
Overall Officials: Chong Bum Chang, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (10):
- South Korea (10):
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do, Gyeonggi-do
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Inha University Hospital, Junggu, Incheon
  - Chung-Ang University Hospital, Dongjak, Seoul
  - Seoul Metropolitan Government-Seoul National University Boramae Medical Center, Dongjak, Seoul
  - Kyung Hee University Hospital at Gangdong, Gangdong, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seocho, Seoul
  - Asan Medical Center, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park TH, Yoon C, Park JH, Lee S, Choi CH, Chang CB, Kim JG. Study protocol for a prospective, randomized controlled confirmatory clinical investigation to evaluate the safety and efficacy of a multidisciplinary digital therapeutics in patients with patellofemoral pain syndrome. Trials. 2025 Sep 1;26(1):328. doi: 10.1186/s13063-025-09030-2. PMID 40890852